CLINICAL TRIAL: NCT04453384
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 (2a and 2b) Study to Evaluate the Safety and Efficacy of XAV-19 in Patients With COVID-19 Induced Moderate Pneumonia
Brief Title: Study to Evaluate the Safety and Efficacy of XAV-19 in Patients With COVID-19 Induced Moderate Pneumonia
Acronym: POLYCOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: BPIfrance (Other); Xenothera SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC20_0230
Record Dates: First submitted 2020-06-22; First posted 2020-07-01 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: SARS Virus
Keywords: SARS-Cov-2; COVID-19; Moderate; pneumonia; antibody
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Lymphoma, Follicular; Pneumonia | interventions — XAV-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Administrations of XAV-19
  * Phase 2a: XAV-19 at 0.5 mg/kg at D1 and D5(Group 1) or at 2 mg/kg at D1 and D5 (Group 2), or at 2 mg/kg at D1 (groupe 3)
  * Phase 2b: Selected dose from Phase 2a : one administration at 2 mg/kg on day1
  Interventions: Drug: XAV-19
- Placebo arm (Placebo Comparator): same administration as treatment arm
  * Phase 2a: two administrations of placebo (day 1 and day 5) for Group 1 and 2, one administration of placebo on day 1 for Group 3
  * Phase 2b: one administration of placebo on day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XAV-19 — Phase 2a: Administration on Day 1 and day 5 for Group1 and 2, Administration on Day 1 for Group 3 Phase 2b: Administration on Day 1
  Arms: Treatment arm
Drug: Placebo — Phase 2a: Administration on Day 1 and day 5 for Group1 and 2, Administration on Day 1 for Group 3 Phase 2b: Administration on Day 1
  Arms: Placebo arm

SUMMARY:
Early inhibition of entry and replication of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a very promising therapeutic approach. Polyclonal neutralizing antibodies offers many advantages such as providing immediate immunity, consequently blunt an early pro-inflammatory pathogenic endogenous antibody response and lack of drug-drug interactions1-3.

Because a suboptimal endogenous early antibody response with regard to SARS-CoV-2 replication in severe cases is observed, neutralising antibody treatment can be very interesting for patient with COVID-19 induced moderate pneumonia4,5. Convalescent plasma to treat infected patients is therefore an interesting therapeutic option currently under evaluation. However, the difficulties of collecting plasma and its safety aspects are not adapted to many patients.

A new polyclonal humanized anti-SARS-CoV2 antibodies (XAV-19) is being developed by Xenothera, which can be administered as intravenous treatment. XAV-19 is a heterologous swine glyco-humanized polyclonal antibody (GH-pAb) raised against the spike protein of SARS-CoV-2, inhibiting infection of ACE-2 positive human cells with SARS-CoV-2. Pharmacokinetic and pharmacodynamic studies have been performed in preclinical models including primates and a First In Human study with another fully representative GH-pAb from Xenothera is ongoing in volunteer patients recipients of a kidney graft. These studies indicated that 5 consecutive administrations of GH-pAbs can be safely performed in humans.

The objective of this 2-steps phase 2 randomized double-blind, placebo-controlled study is 1) to define the optimal and safety XAV-19 dose to administrate in patients with COVID-19 induced moderate pneumonia ; 2) to show the clinical benefit of selected dose of XAV-19 when administered to patients with COVID-19 induced moderate pneumonia.

DETAILED DESCRIPTION:
For the first set of statistical analyses, to allow early reporting of primary and secondary endpoints at D15, the blind will be partially broken once all patients have completed Day 29. Except for statisticians, only the principal investigator and the scientific coordinator will have access to the full data set for the analysis of the primary and secondary endpoints up to day 29. The database will be partially locked (with all data up to day 29) as neither monitors nor investigators will be informed of the unblinding until the final data for day 60 is completed and the final database is locked.

ELIGIBILITY:
Phase 2a:

Inclusion Criteria:

1. Willing and able to provide written informed consent prior to performing study procedures
2. Male or female ≥ 18 years and ≤ 85 years
3. Hospitalized for COVID-19
4. Positive SARS-CoV-2 RT-PCR in any body specimen (nasopharynx, saliva, sputum) ≤ 10 days before enrolment
5. Evidence of pulmonary involvement (on lung examination [rales/crackles] and/or chest-imaging [Chest X-ray or computed tomography])
6. Requiring O2 supplement ≤ 6L/min at screening
7. Requiring O2 supplementation with SpO2 ≥ 94% on O2 therapy at screening
8. First onset of COVID-19 symptoms ≤ 10 days, among fever and/or chills, headache, myalgias, cough, shortness of breath, whichever as occurred fist
9. WOCBP must have a negative urinary pregnancy test the day of inclusion
10. All sexually active male subjects must agree to use an adequate method of contraception throughout the study period and for 90 days after the last dose of study drug and agree to no sperm donation until the end of the study, or for 90 days after the last dose of XAV-19, whichever is longer
11. Patients with French social security

Exclusion Criteria:

1. Evidence of multiorgan failure (severe COVID-19)
2. Mechanically ventilated (including ECMO)
3. Receipt of immunoglobulins or any blood products in the past 30 days
4. Psychiatric or cognitive illness or recreational drug/alcohol use that in the opinion of the investigator, would affect subject safety and/or compliance
5. End-stage renal disease (eGFR < 15 ml/min/1,73 m2)
6. Child-Pugh C stage liver cirrhosis
7. Decompensated cardiac insufficiency
8. History of active drug abuse
9. Known allergy, hypersensitivity, or intolerance to the study drug, or to any of its components
10. Females of childbearing potential without contraceptive method, or with positive pregnancy test, breastfeeding, or planning to become pregnant during the study period
11. Current documented and uncontrolled bacterial infection.
12. Prior severe (grade 3) allergic reactions to plasma transfusion
13. Patient participating in another interventional clinical trial
14. Life expectancy estimated to be less than 6 months
15. Patient under guardianship or trusteeship

Phase 2b:

Inclusion criteria:

1. Willing and able to provide written informed consent prior to performing study procedures
2. Male or female ≥ 18 years
3. Hospitalized for COVID-19
4. Documentation of SARS-Cov-2 infection before enrolment, by positive SARS-CoV-2 RT-PCR or antigen in any body specimen (nasopharynx, oropharynx, saliva, sputum, bronchoalveolar lavage …) before enrolment
5. Evidence of pulmonary involvement (on lung examination [rales/crackles] and/or chestimaging [Chest X-ray or computed tomography])
6. Requiring O2 supplement ≤ 6L/min at screening
7. Requiring O2 supplementation with SpO2 ≥ 92% on O2 therapy at screening (or ≥ 90

   % if chronic obstructive pulmonary disease)
8. First onset of COVID-19 symptoms ≤ 14 days, among fever and/or chills, headache, myalgias, cough, shortness of breath, whichever as occurred fist (other symptoms such as asthenia not to be considered in this list)
9. WOCBP must have a negative urinary pregnancy test the day of inclusion
10. All sexually active male subjects must agree to use an adequate method of contraception throughout the study period and for 90 days after the last dose of study drug and agree to no sperm donation until the end of the study, or for 90 days after the last dose of XAV-19, whichever is longer
11. Patients with French social security

Exclusion criteria:

1. Evidence of multiorgan failure (severe COVID-19)
2. Mechanically ventilated (including ECMO)
3. Receipt of immunoglobulins or any blood products in the past 30 days
4. Psychiatric or cognitive illness or recreational drug/alcohol use that in the opinion of the investigator, would affect subject safety and/or compliance
5. End-stage renal disease (eGFR < 15 ml/min/1,73 m2)
6. Child-Pugh C stage liver cirrhosis
7. Decompensated cardiac insufficiency
8. Known allergy, hypersensitivity, or intolerance to the study drug, or to any of its components
9. Females of childbearing potential without contraceptive method, or with positive pregnancy test, breastfeeding, or planning to become pregnant during the study period
10. Current documented and uncontrolled bacterial infection.
11. Prior severe (grade 3) allergic reactions to plasma transfusion
12. Patient participating in another interventional clinical trial
13. Life expectancy estimated to be less than 6 months
14. Patient under guardianship or trusteeship
15. Patient already included
16. Prior hospitalisation in intensive care unit for the current covid-19 episode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Phase 2a: XAV-19 antibody titers | Day 8
  The primary endpoint is measurement of the antibody titer XAV-19 in all treated patients and in all patients in the placebo group at Day 8
Phase 2a: Adverse events of XAV-19 | Day 29
  Adverse events of XAV-19 between the two groups of treated patients and vs. placebo over 29 days
Phase 2b: To evaluate the efficacy of XAV-19 + standard-of-care (Soc) therapy compared with placebo + Soc therapy for treatment of COVID-19 assessed by the proportion of patients who die or develop respiratory failure between baseline and Day 15. | Day 15
  Efficacy is defined by the proportion of patients who died or develop respiratory failure, as defined by the requirement of noninvasive ventilation, high-flow oxygen devices, invasive mechanical ventilation (corresponding to a score of 5 or more on the WHO 8 point ordinal scale) or by an increase of the required O2 supplement (more or equals to 10 L/minutes with a non-rebreather mask (oxygen mask with reservoir bag)

SECONDARY OUTCOMES:
Phase 2a: Pharmacokinetic analysis | Day 1 (pre-dose, post-dose), at Day 5 (pre-dose, post-dose), Day 8, Day 15, and Day 29
  XAV-19 Antibody titer over the time
Phase 2a: Antibody titer between the two groups | day 15
  The antibody titer of XAV-19 measurements in Group 1 treated patients and Group 2 treated patients
Phase 2a: Supplemental oxygen | Day 1 to Day 29
  Duration of supplemental oxygen
Phase 2a: Evaluation of Transfer to intensive care | Day 1 to Day 29
  Transfer to intensive care unit with need for invasive mechanical ventilation or high flow oxygen
Phase 2a: Normalization of Fever | Day 1 to Day 29
  Normalization of fever ≥ 24 hours: clinical assessment every day from Day 1 to Day 14. Evaluation to be performed between 8 and 12 am, Day X evaluation will consider the higher value during Day X-1
Phase 2a: Biomarkers | Day 1 to Day 29
  Biomarkers : CRP, Ferritin
Phase 2a: Hospital length of stay | Day 1 to Day 29
  Evaluation of Hospital length of stay
Phase 2b: Efficacy of XAV-19 | Day 8 and Day 29
  Proportion of patients who die, develop respiratory failure, as defined by the requirement of noninvasive ventilation, high-flow oxygen devices or invasive mechanical ventilation at Day 8 and D29
Phase 2b: Clinical severity | Day 3, Day 5, Day 8, Day15 and Day 29
  a) National Early Warning Score (NEWS) assessed while hospitalized and on Day 15 and Day 29
Phase 2b: Clinical severity | Day 29
  b) Clinical status using the 8-point ordinal scale assessed daily until Day 29
Phase 2b: Clinical severity : Improvement of clinical and biological parameters | Day15, and Day 29
  c) Temperature and blood analysis between baseline and Day 15, and Day 29
Phase 2b: Clinical severity : Oxygenation | 29 Days
  d) Days of oxygen therapy over 29 days PaO2 / FiO2 at baseline, Day 5, Day 8, Day 15, Day 29 if available
Phase 2b: Clinical severity : Non-invasive ventilation, high-flow oxygen | 29 Days
  e) e) Days of non-invasive ventilation or high flow oxygen (if applicable) up to Day 29
Phase 2b: Clinical severity : Invasive mechanical ventilation / Extra Corporeal Membrane Oxygenation (ECMO) | 29 Days
  f) Days of invasive mechanical ventilation/ECMO (if applicable) up to Day 29
Phase 2b: Clinical severity : Transfer in ICU by Day 29 | 29 Days
  g) Transfer in ICU
Phase 2b: Clinical severity : Hospitalization | 60 Days
  h) Hospital length of stay (in days)
Phase 2b: Clinical severity : Mortality | 60 Days
  i) All-cause mortality evaluated between baseline and Day 15 and between baseline and at Day 29 and at Day 60
Phase 2b: Clinical severity : Thrombotic events | 60 Days
  j) Thrombotic events (peripheral venous, pulmonary, arterial)
Phase 2b: mortality | 29 Days
  k) All cause mortality
Phase 2b: safety | 29 days and 60 days
  Occurrence of all suspected XAV-19 related adverse effects or Incidence of serious adverse events
Phase 2b: safety of Study drug infusion | 29 days and 60 days
  Study drug discontinuation or temporary suspension of infusion
Phase 2b: safety : study drug discontinuation | 29 days and 60 days
  Proportion of participants with treatment emergent adverse events leading to study drug discontinuation
Phase 2b: safety : major or opportunistic bacterial or fungal infections | 29 days and 60 days
  Incidence of major or opportunistic bacterial or fungal infections
Phase 2b: safety : hypersensitivity reactions and infusion reactions | 29 days and 60 days
  Incidence of hypersensitivity reactions and infusion reactions
Phase 2b: safety : biological parameters | 29 days and 60 days
  White cell count, hemoglobin, platelets, creatinine, ALT, AST, on D1, D3, D5, D8, D15 and D29
Phase 2b: Exploratory analysis : qualitative and quantitative SARS-CoV-2 status | Day 1, Day 8, Day 15 and Day 29
  SARS-CoV-2 status (positive or negative and quantitatively, including variant information by sequencing) over time (D1, D8, D15, and D29)
Phase 2b: Exploratory analysis : SARS-CoV-2 status viral load | Day 1, Day 8, Day 15 and Day 29
  SARS-CoV-2 status viral load over time (D1, D8, D15, and D29)

OTHER OUTCOMES:
Phase 2b : Pharmacokinetic Study | Day 1, Day 3, Day 5, Day 8, Day 15 and Day 29
  Pharmacokinetic analysis correspond to antibody titer measurements at Day 1 (pre-dose, post-dose), Day 3, Day 5, Day 8, Day 15, and Day 29
Phase 2b : Immunomonitoring Study | Day 1, Day 3, Day 5, Day 8, Day 15 and Day 29
  The endpoints encompass the following analysis:
  * Spike/ACE2 neutralizing antibody titers: D1 (pre-, post dose), D3, D5, D8, D15 and D29
  * Lymphocytes sub-population: D1, D3, D5, D8 and D15
  * Transcriptomic analyses: D1, D3, D5, D8 and D15
  * Cytokines: D1, D3, D5, D8 and D15
Phase 2b : Terminal ancillary Study (20 additional patients receiving a fixed dose of 150mg of XAV-19 : | Day 1, Day 3, Day 5, Day 8, Day 15 and Day 29
  * to compare pharmacokinetic parameters in patients receiving a fixed dose of 150mg with patients receiving 2mg/Kg of XAV-19 (master phase 2b), in order to confirm that the exposure and variability are similar
  * to compare the effects of neutralizing antibodies use on virus-induced immune response on longitudinal follow-up, and targets for "immuno-monitoring"
  * to investigate the immunogenicity of COVID-19 during treatment with XAV19 in patients receiving a fixed dose of 150mg with patients receiving 2mg/Kg of XAV-19

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Gaborit, Principal Investigator — Nantes University Hospital
Locations (34):
- France (32):
  - CHU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - Hôpital Privé d'Antony, Antony
  - CH Avignon, Avignon
  - CH de la Côte Basque, Bayonne
  - APHP - Hôpital Avicennes, Bobigny
  - CHU Caen, Caen
  - CH Métropole Savoie, Chambéry
  - CH Colmar, Colmar
  - CH Sud Francilien, Corbeil-Essonnes
  - CHD Vendée, La Roche-sur-Yon
  - CH de La Rochelle, La Rochelle
  - CH Le Mans, Le Mans
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - Hospices Civils Lyon, Lyon
  - CH de Mont de Marzan, Mont-de-Marsan
  - GHR Mulhouse Sud-Alsace, Mulhouse
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU Nîmes, Nîmes
  - CHR Orléans La Source, Orléans
  - APHP - Hôpital Tenon, Paris
  - Hôpital Saint Antoine, Paris
  - CH René Dubos, Pontoise
  - CH Cornouaille, Quimper
  - CHU Reims, Reims
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - CHU Strasbourg, Strasbourg
  - Hôpital FOCH, Suresnes
  - CHRU Nancy, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique, Vannes
- CHU Martinique, Fort-de-France, Martinique
- CHU La Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimber C, Valk SJ, Chai KL, Piechotta V, Iannizzi C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Hyperimmune immunoglobulin for people with COVID-19. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD015167. doi: 10.1002/14651858.CD015167.pub2. PMID 36700518
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Gaborit B, Dailly E, Vanhove B, Josien R, Lacombe K, Dubee V, Ferre V, Brouard S, Ader F, Vibet MA, Le Thuaut A, Danger R, Flet L, Omnes A, Berly L, Chiffoleau A, Jobert A, Duvaux O, Raffi F; POLYCOR Trial Group. Pharmacokinetics and Safety of XAV-19, a Swine Glyco-humanized Polyclonal Anti-SARS-CoV-2 Antibody, for COVID-19-Related Moderate Pneumonia: a Randomized, Double-Blind, Placebo-Controlled, Phase IIa Study. Antimicrob Agents Chemother. 2021 Aug 17;65(9):e0123721. doi: 10.1128/AAC.01237-21. Epub 2021 Aug 17. PMID 34181475
- [Derived] Gaborit B, Vanhove B, Vibet MA, Le Thuaut A, Lacombe K, Dubee V, Ader F, Ferre V, Vicaut E, Orain J, Le Bras M, Omnes A, Berly L, Jobert A, Morineau-Le Houssine P, Botturi K, Josien R, Flet L, Degauque N, Brouard S, Duvaux O, Poinas A, Raffi F; POLYCOR study group. Evaluation of the safety and efficacy of XAV-19 in patients with COVID-19-induced moderate pneumonia: study protocol for a randomized, double-blinded, placebo-controlled phase 2 (2a and 2b) trial. Trials. 2021 Mar 9;22(1):199. doi: 10.1186/s13063-021-05132-9. PMID 33750432